CLINICAL TRIAL: NCT06405971
Title: Metformin in Patients with Unruptured Vertebrobasilar Dissecting Aneurysms: a Prospective, Randomized Study (METTLE)
Brief Title: Metformin in Patients with Unruptured Vertebrobasilar Dissecting Aneurysms (METTLE)
Acronym: METTLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ming Lv (Other)
Responsible Party: Sponsor-Investigator, Ming Lv, Principal Investigator, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ming Lv
Record Dates: First submitted 2024-04-28; First posted 2024-05-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Dissecting Aneurysm of Cerebral Artery
Keywords: Vertebrobasilar dissecting aneurysms; Metformin; High-resolution vessel wall imaging; Inflammatory reaction
MeSH Terms: conditions — Inflammation | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Simple randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To ensure the reliability of the research results, a study committee consisting of 5 members will be formed. The committee comprised a 2-member data safety monitoring committee and a 3-member clinical event review committee. These committee members were blinded to the treatment group assignments. Any disagreements were resolved by a third member of the clinical events adjudication committee. All five committee members reviewed and resolved any discrepancies through consensus.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug Group (Experimental): Patients in the drug group were given one oral tablet of metformin hydrochloride enteric capsule each day after breakfast and dinner at a dose of 250 mg per tablet.
  Interventions: Drug: Metformin
- Placebo group (Placebo Comparator): Patients in the placebo group were given one oral tablet of placebo (capsule filled with corn starch) each day after breakfast and dinner at a dose of 250 mg per tablet.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Patients in the drug group took one tablet of metformin hydrochloride enteric capsule orally each day after breakfast and dinner, and the dose of each tablet was 250mg.

SUMMARY:
Vertebrobasilar dissecting aneurysms (VBDAs) are one of the most important causes of stroke in young and middle-aged people, and the natural history of VBDAs is complex and varied, often leading to high rates of disability and mortality. For some patients with VBDAs who are not suitable for surgical entrapment and intervention, pharmacologic therapy may be used to slow the progression of VBDAs. Metformin (MET) has been shown to act as an anti-inflammatory, anti-oxidative stress and improve vascular endothelial function by inhibiting smooth muscle cell phenotypic transformation, proliferation, migration and apoptosis, thereby reducing the incidence of intracranial aneurysms and rupture rates, and MET may be a suitable candidate. Inflammatory response plays an important role in the occurrence, development and rupture of VBDAs. Inflammatory response in the aneurysm wall can cause endothelial and smooth muscle cell injury and apoptosis, leading to degenerative changes in the vessel wall and increasing the risk of rupture of VBDAs. High-resolution magnetic resonance vessel wall imaging (HR-VWI), which can clearly show the structure of the vessel wall and reflect the active degree of inflammatory reaction in the aneurysm wall, has been widely used in the assessment of intracranial aneurysm instability. In this study, we propose to conduct a multicenter, prospective, randomized study to investigate whether MET reduces the degree of aneurysm wall inflammatory response in VBDAs by performing HR-VWI scans in patients with VBDAs and obtaining quantitative parameters reflecting the inflammatory response of the aneurysm wall.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years, gender is not limited;
2. Patients with previously untreated, unruptured stable VBDAs clearly diagnosed by DSA, CTA or MRA;
3. Patients with aneurysm wall enhancement as shown by HR-VWI of 3.0T high field strength MRI whole body scanner at Tsinghua University;
4. Baseline mRS score ≤2;
5. Patients voluntarily participated in this study and signed an informed consent form.

Exclusion Criteria:

1. Patients with aneurysms located in non-vertebral basilar artery sites (mainly referring to bifurcation saccular aneurysms);
2. Patients with combined diabetes or its complications;
3. Patients who are allergic to any components in MET;
4. Pregnant and lactating female patients;
5. Patients with other immune diseases in combination, patients taking immunosuppressants or anti-inflammatory drugs (such as long-term use of aspirin, statin, hormones and other drugs);
6. Target aneurysm-related symptoms were severe at the time of diagnosis, and the mRS score was ≥3;
7. VBDAs have received interventional or surgical treatment;
8. Those with severe allergy to the contrast agent gadolinium terlumate glucosamine (Gd-DTPA) (skin rash not counted);
9. Those with severe renal disease resulting in renal insufficiency (glomerular filtration rate <30ml/(min·1.73m2));
10. Patients with metal implants in the body (e.g., cardiac stents, cardiac prosthetic valves, pacemakers, metal joints, steel plates, non-removable metal dentures, etc.);
11. Patients known to suffer from dementia or psychiatric disorders and claustrophobia who are unable to complete the magnetic resonance examination;
12. Patients with other serious diseases combined at the time of diagnosis and with an expected survival time of less than 1 year;
13. Patients who are participating in clinical trials of other drugs or devices.
14. Other conditions judged by the investigator to exist that are unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
3-dimensional wall enhancement volume rate (3D-WEVR) | 6 months after taking the drug
  Changes in the degree of wall enhancement of VBDAs at the time of patient enrollment and after 6 months of oral drug administration were measured by HR-VWI, i.e., the quantitative wall enhancement parameters 3D-WEVR was compared between the drug group and the placebo group at the end of the 6-month treatment period. The unit of 3D-WEVR is percentage (%).

SECONDARY OUTCOMES:
Morphological changes in VBDAs | 6 months after taking the drug
  change in the maximum diameter of the aneurysm by ≥1 mm or the presence of a daughter aneurysm was defined as a morphologic change
Characteristic changes in the internal lumen of VBDAs | 6 months after taking the drug
  change of intramural hematoma by ≥1 mm or disappearance of false lumen defined as characteristic changes in the internal lumen
Changes in C-reactive protein | 6 months after taking the drug
  The unit of C-reactive protein is mg/dL.
changes in serum inflammatory markers | 6 months after taking the drug
  e.g., IL-1β, IL-2R, IL-6, IL-8, IL-10, TNF-α. The unit of serum inflammatory markers is pg/ml.
changes in serum inflammatory markers | 6 months after taking the drug
  e.g., MMP-3, MMP-9. The unit of serum inflammatory markers is ng/ml.
Proportion of patients with VBDAs who developed cerebral infarction, transient ischemic attack, cerebral hemorrhage, and symptoms of compression in the drug and placebo groups were recorded | 6 months after taking the drug
  To record patients with VBDAs who developed cerebral infarction, transient ischemic attack, cerebral hemorrhage, and pressure symptoms in the drug and placebo groups, and to clarify whether MET suppresses ischemic events, hemorrhagic events, and pressure-occupying events (defined as ischemic events, hemorrhagic events, and pressure-occupying events if the patient's mRS scores are increased and associated with a target aneurysm)
Wall enhancement index (WEI) | 6 months after taking the drug
  Changes in the degree of wall enhancement of VBDAs at the time of patient enrollment and after 6 months of oral drug administration were measured by HR-VWI, i.e., the quantitative wall enhancement parameters WEI was compared between the drug group and the placebo group at the end of the 6-month treatment period. Quantitative parameter WEI has no units.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Schievink WI. Spontaneous dissection of the carotid and vertebral arteries. N Engl J Med. 2001 Mar 22;344(12):898-906. doi: 10.1056/NEJM200103223441206. No abstract available. PMID 11259724
- [Background] Debette S, Compter A, Labeyrie MA, Uyttenboogaart M, Metso TM, Majersik JJ, Goeggel-Simonetti B, Engelter ST, Pezzini A, Bijlenga P, Southerland AM, Naggara O, Bejot Y, Cole JW, Ducros A, Giacalone G, Schilling S, Reiner P, Sarikaya H, Welleweerd JC, Kappelle LJ, de Borst GJ, Bonati LH, Jung S, Thijs V, Martin JJ, Brandt T, Grond-Ginsbach C, Kloss M, Mizutani T, Minematsu K, Meschia JF, Pereira VM, Bersano A, Touze E, Lyrer PA, Leys D, Chabriat H, Markus HS, Worrall BB, Chabrier S, Baumgartner R, Stapf C, Tatlisumak T, Arnold M, Bousser MG. Epidemiology, pathophysiology, diagnosis, and management of intracranial artery dissection. Lancet Neurol. 2015 Jun;14(6):640-54. doi: 10.1016/S1474-4422(15)00009-5. PMID 25987283
- [Background] Sikkema T, Uyttenboogaart M, Eshghi O, De Keyser J, Brouns R, van Dijk JM, Luijckx GJ. Intracranial artery dissection. Eur J Neurol. 2014 Jun;21(6):820-6. doi: 10.1111/ene.12384. Epub 2014 Feb 22. PMID 24824740
- [Background] Quan K, Song J, Yang Z, Wang D, An Q, Huang L, Liu P, Li P, Tian Y, Zhou L, Zhu W. Validation of Wall Enhancement as a New Imaging Biomarker of Unruptured Cerebral Aneurysm. Stroke. 2019 Jun;50(6):1570-1573. doi: 10.1161/STROKEAHA.118.024195. Epub 2019 Apr 30. PMID 31035900
- [Background] Larsen N, von der Brelie C, Trick D, Riedel CH, Lindner T, Madjidyar J, Jansen O, Synowitz M, Fluh C. Vessel Wall Enhancement in Unruptured Intracranial Aneurysms: An Indicator for Higher Risk of Rupture? High-Resolution MR Imaging and Correlated Histologic Findings. AJNR Am J Neuroradiol. 2018 Sep;39(9):1617-1621. doi: 10.3174/ajnr.A5731. Epub 2018 Jul 19. PMID 30026386
- [Background] Lv N, Karmonik C, Chen S, Wang X, Fang Y, Huang Q, Liu J. Wall Enhancement, Hemodynamics, and Morphology in Unruptured Intracranial Aneurysms with High Rupture Risk. Transl Stroke Res. 2020 Oct;11(5):882-889. doi: 10.1007/s12975-020-00782-4. Epub 2020 Jan 20. PMID 31960286
- [Background] Etminan N, Rinkel GJ. Unruptured intracranial aneurysms: development, rupture and preventive management. Nat Rev Neurol. 2016 Dec;12(12):699-713. doi: 10.1038/nrneurol.2016.150. Epub 2016 Nov 3. PMID 27808265
- [Background] Shimonaga K, Matsushige T, Ishii D, Sakamoto S, Hosogai M, Kawasumi T, Kaneko M, Ono C, Kurisu K. Clinicopathological Insights From Vessel Wall Imaging of Unruptured Intracranial Aneurysms. Stroke. 2018 Oct;49(10):2516-2519. doi: 10.1161/STROKEAHA.118.021819. PMID 30355091
- [Background] He J, Li N, Fan Y, Zhao X, Liu C, Hu X. Metformin Inhibits Abdominal Aortic Aneurysm Formation through the Activation of the AMPK/mTOR Signaling Pathway. J Vasc Res. 2021;58(3):148-158. doi: 10.1159/000513465. Epub 2021 Feb 18. PMID 33601368
- [Background] Maruthur NM, Tseng E, Hutfless S, Wilson LM, Suarez-Cuervo C, Berger Z, Chu Y, Iyoha E, Segal JB, Bolen S. Diabetes Medications as Monotherapy or Metformin-Based Combination Therapy for Type 2 Diabetes: A Systematic Review and Meta-analysis. Ann Intern Med. 2016 Jun 7;164(11):740-51. doi: 10.7326/M15-2650. Epub 2016 Apr 19. PMID 27088241
- [Background] Rena G, Hardie DG, Pearson ER. The mechanisms of action of metformin. Diabetologia. 2017 Sep;60(9):1577-1585. doi: 10.1007/s00125-017-4342-z. Epub 2017 Aug 3. PMID 28776086
- [Background] Cameron AR, Morrison VL, Levin D, Mohan M, Forteath C, Beall C, McNeilly AD, Balfour DJ, Savinko T, Wong AK, Viollet B, Sakamoto K, Fagerholm SC, Foretz M, Lang CC, Rena G. Anti-Inflammatory Effects of Metformin Irrespective of Diabetes Status. Circ Res. 2016 Aug 19;119(5):652-65. doi: 10.1161/CIRCRESAHA.116.308445. Epub 2016 Jul 14. PMID 27418629
- [Background] Li S, Shi Y, Liu P, Song Y, Liu Y, Ying L, Quan K, Yu G, Fan Z, Zhu W. Metformin inhibits intracranial aneurysm formation and progression by regulating vascular smooth muscle cell phenotype switching via the AMPK/ACC pathway. J Neuroinflammation. 2020 Jun 16;17(1):191. doi: 10.1186/s12974-020-01868-4. PMID 32546267
- [Derived] Dong L, Xu Z, Li Y, Wei D, Lin J, Wang C, Chen H, Lv M. Metformin for the treatment of unruptured vertebrobasilar dissecting aneurysm (METTLE): study protocol for a double-blinded randomised controlled trial. Trials. 2025 Dec 6;27(1):27. doi: 10.1186/s13063-025-09348-x. PMID 41351119